CLINICAL TRIAL: NCT03125408
Title: Clinical Utility of the DxN HCV Assay as an Aid in the Management of HCV-Infected Individuals Undergoing Antiviral Therapy
Brief Title: Clinical Performance Evaluation of DxN HCV Assay
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HCV 2.7.3.001
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen plasma samples are retained for this study and possible future studies.
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- chronic HCV Infected patients: chronic HCV patients who will undergo standard of care FDA approved antiviral therapy to treat genotype 1,2, or 3 infections and will have blood drawn at various time points and tested using the DxN HCV Assay. Study is observational and results will not be used to manage patient care.
  Interventions: Diagnostic Test: HCV Assay

INTERVENTIONS:
Diagnostic Test: HCV Assay — Molecular diagnostic test to detect Hepatitus C
  Other Names: DxN HCV Assay

SUMMARY:
The DxN Hepatitis C Virus (HCV) Assay is an in vitro diagnostic assay intended as an aid in the management of of HCV-infected individuals undergoing antiviral therapy. The purpose of the study is to establish the clinical performance of the DxN HCV Assay for plasma samples in the intended use population.

DETAILED DESCRIPTION:
Same as brief

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has measurable HCV-RNA at baseline (prior to treatment start)
* Subject is genotype 2 or 3 and plans to undergo treatment with Peginterferon (PEG) plus Ribavirin (RBV) or Sofosbuvir (SOF) plus RIB
* Subject is genotype 1 and plans to undergo treatment with Telaprevir (TEL) or SOF plus PEG+RBV or, SOF plus Ledipasivr (LED)
* Subject is able to under information given, and willing and able to voluntarily give their consent to participate in study including signing consent form.

Exclusion Criteria:

* Co-infection with HIV or Hepatitis B (HBV)
* Prior participation in study
* Current participation in an investigation drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older with chronic HCV who will undergo antiviral therapy to treat genotype 1,2 or 3 infections.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-05-02; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | Up to 9 months
  Defined as unquantifiable HCV Viral load after discontinuation of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- SC Liver Research Consortium, Duluth, Georgia, United States

IPD SHARING:
Plan to Share IPD: No